CLINICAL TRIAL: NCT07127770
Title: A Phase 1, Open-label, Fixed Sequence, 2-period Study in Healthy Adult Male Participants to Assess the Mass Balance, Absolute Bioavailability, Fraction Absorbed, and Pharmacokinetics of [ 14C]PF-07104091
Brief Title: A Study to Understand How the Body Processes [14C]PF-07104091 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C4161006; 2024-518696-65-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-07-01; First posted 2025-08-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adults
Keywords: Pharmacokinetics; Healthy Volunteers; Biological Availability; Absorption; Elimination; Distribution; ADME; Bioavailability; Radiolabeled; Metabolic Profile; Renal Elimination; Mass Balance; Small molecule; Absolute Bioavailability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A; Period 1 (Experimental): Single oral dose of 14C-labeled PF-07104091 administered under fed conditions.
  Interventions: Drug: PF-07104091
- Regimen B; Period 2 (Experimental): Single oral dose of unlabeled PF-07104091 administered under fed conditions followed by an intravenous (IV) infusion of PF-07104091 containing a microdose of 14C-labeled PF-07104091.
  Interventions: Drug: PF-07104091

INTERVENTIONS:
Drug: PF-07104091 — Cyclin-dependent kinase-2 inhibitor

SUMMARY:
The purpose of this study is to learn how the body processes the study medicine PF-07104091.

The study is seeking participants who are:

- Healthy male aged 18 to 65 years of age

Participants in the study will receive 14C-labeled PF-07104091 by mouth after a meal. After 14 days, the participants will receive PF-07104091 by mouth (after a meal) followed by IV fusion (given directly into a vein) of microdose [14C]PF-07104091.

The study will help understand how the body processes study medicine PF-07104091 and how the medicine is changed and removed from the body after you take it. This study will also help to understand how much PF-07104901 is taken up into the blood.

Participants will remain in the study clinic for a maximum of 23 days and will have one follow-up contact.

ELIGIBILITY:
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and standard 12-lead ECGs.
* Body mass index (BMI) of 17.5-32.0 kg/m2 inclusive and a total body weight >50 kg (110 lb)
* Evidence of a personally signed and dated Informed Consent Document (ICD) indicating that the participant has been informed of all pertinent aspects of the study.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and standard 12-lead ECGs
Enrollment: 9 (Actual)
Dates: Start 2025-08-28 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Total Radiocarbon (14c) excreted in urine | From Predose up to 14 days post dose of period 1 and 2
  Percentage of 14C excreted in urine following 14C PF-07104091 single dose administration will be determined as: (Total 14C urine/ 14C dose administered) *100 where, 14C dose was administered dose of 14C PF-07104091.
Percentage of Total Radiocarbon (14c) excreted in feces | From Predose up to 14 days post dose of period 1 (and if applicable for Period 2)
  Percentage of 14C excreted in feces following 14C PF-07104091 single dose administration will be determined as: (Total 14C feces/ 14C dose administered) *100 where, 14C dose was administered dose of 14C PF-07104091.
Percentage of Total Radiocarbon (14c) excreted in vomitus (if applicable) | From Predose up to 14 days post dose of period 1 only
  Percentage of 14C excreted in vomitus (if applicable) following 14C PF-07104091 single dose administration will be determined as: (Total 14C vomitus/ 14C dose administered) *100 where, 14C dose was administered dose of 14C PF-07104091.
Cumulative Percent Recovery of Total Radiocarbon (14C) | From Predose up to 14 days post dose of period 1 only
  Percentage recovery of total radioactivity (14C) in urine, feces, and vomitus (If applicable) was determined based on total administered dose.
Percentage of Metabolite Detected in Plasma After Oral Administration of PF-07104091 | From Predose to 14 days post dose of period 1
  The percentage of major metabolites detected in plasma after oral administration of PF-07104091
Percentage of Metabolite Detected in Urine After Oral Administration of PF-07104091 | From Predose to 14 days post dose of period 1
  The percentage of major metabolites detected in urine after oral administration of PF-07104091
Percentage of Metabolite Detected in Feces After Oral Administration of PF-07104091 | From Predose to 14 days post dose of period 1
  The percentage of major metabolites detected in feces after oral administration of PF-07104091

SECONDARY OUTCOMES:
Oral Absolute Bioavailability | From Predose up to 14 days post dose, period 2 only.
  Dose normalized AUCinf (AUCinf[dn]) will be calculated as AUCinf/Dose, where AUCinf is the area under the plasma concentration-time profile from time 0 extrapolated to infinite time. Absolute oral bioavailability is defined as the ratio of geometric mean of AUCinf(dn) following orally administered PF-07104091 (i.e., unlabeled PF-07104091) to AUCinf(dn) following intravenously administered [14C]PF-07104091 in period 2.
Fraction of PF-07104091 Dose Absorbed (Fa) | From Predose up to 14 days post dose
  Fraction of dose absorbed (Fa) will be estimated as the ratio of total or partial radioactivity (dose normalized) excreted into the urine (from time 0 to the time of last measurable concentration) following oral and IV administration of [14C]PF-07104091 microtracer dose in Period 1 and 2, respectively.
Number of Participants with Clinically Significant Abnormalities in Laboratory Parameters | From baseline up to 35 days after the last dose of study intervention (up to Day 36)
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | From baseline up to 35 days after the last dose of study intervention (up to Day 36)
Number of Participants With Clinically Significant Abnormalities in Vital Signs | From baseline up to 35 days after the last dose of study intervention (up to Day 36)
Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities | From baseline up to 35 days after the last dose of study intervention (up to Day 36)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4161006